CLINICAL TRIAL: NCT05960149
Title: Evaluation of the Effect of Intraoperative Indocyanine Green Use on Erectile Function and Surgical Margin Positivity in Patients Undergoing Nerve-Sparing Robot-Assisted Laparoscopic Radical Prostatectomy
Brief Title: Use of Indocyanine Green in Robotic Prostate Surgeries
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Araz Musaev, Principal İnvesitgator, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A01062021Z
Record Dates: First submitted 2023-05-31; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Prostate Cancer Adenocarcinoma; Erectile Dysfunction Following Radical Prostatectomy
Keywords: erectile dysfunction and indocyanine green; radical prostatectomy and indocyanine green
MeSH Terms: conditions — Erectile Dysfunction | interventions — Indocyanine Green

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group using Indocyanine Green (Experimental): Performing nerve-sparing robot-assisted laparoscopic radical prostatectomy by IV injecting of Indocyanine Green
  Interventions: Drug: using Indocyanine Green
- The Indocyanine Green -unused group (Experimental): Nerve-sparing robot-assisted laparoscopic radical prostatectomy without the use of Indocyanine Green
  Interventions: Procedure: Nerve-sparing robot-assisted laparoscopic radical prostatectomy

INTERVENTIONS:
Drug: using Indocyanine Green — Nerve-sparing robot-assisted laparoscopic radical prostatectomy using Indocyanine Green
  Other Names: IV Indocyanine Green injection
  Arms: Group using Indocyanine Green
Procedure: Nerve-sparing robot-assisted laparoscopic radical prostatectomy — Nerve-sparing robot-assisted laparoscopic radical prostatectomy without the use of Indocyanine Green
  Arms: The Indocyanine Green -unused group

SUMMARY:
Imaging of the vascular nerve bundle using Indocyanine Green

DETAILED DESCRIPTION:
Comparison of erectile function and surgical margin positivity after nerve-sparing robot-assisted laparoscopic radical prostatectomy surgery performed by imaging the vascular nerve bundle using Indocyanine Green with the results after nerve-sparing robot-assisted laparoscopic radical prostatectomy surgery without Indocyanine Green

ELIGIBILITY:
Inclusion Criteria:

* Patients with low-intermediate risk prostate cancer

Exclusion Criteria:

* Patients high risk prostate cancer

Max Age: 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-07-30 (Estimated); Primary Completion 2025-12-03 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of erectile function. | up to 12 months
  Evaluation of erectile function after Nerve Sparing Robot Assisted Laparoscopic Radical Prostatectomy with and without the application of Indocyanine Green.Evaluation of surgical margin positivity after Nerve Sparing Robot Assisted Laparoscopic Radical Prostatectomy with and without the application of Indocyanine Green.
  Both groups will evaluate their erectile function by completing the preoperative International Index of Erectile Function Every groups of participants will fill the International Index of Erectile Function -5 again after surgery in 3. -6. -9. -12 months.
  The possible scores for the International Index of Erectile Function- 5 range from 0 to 30, and Erectile disfonction is classified into five categories based on the scores: severe (0-10), moderate (11-16), mild to moderate (17-21), mild (22-25), and no erectile disfonction (26-30).
Evaluation of surgical margin positivity | Up to 12 months
  Postoperative surgical margin positivity will be compared in both groups according to the results of the postoperative pathology report. Surgical margin positivity in both groups will be evaluated as a percentage and it will be evaluated whether there is a significant difference between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Araz Musaev, Principal Investigator — Ankara Universitry

IPD SHARING:
Plan to Share IPD: No